CLINICAL TRIAL: NCT03735459
Title: Impact of an Atopic Dermatitis Education, Reminder, and Accountability Program on Patient Adherence to Treatment and Outcome of Atopic Dermatitis
Brief Title: Eczema Reminder and Accountability Program
Acronym: ERAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Allergy (Unknown)
Responsible Party: Principal Investigator, Vince Wu, McMaster Co-op Student, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERAP
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Treatment adherence and compliance
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient reminder (Experimental): Patient Oriented SCORAD (PO-SCORAD): Assess severity of eczema.
  Adherence Questionnaire (AQ): Assess adherence to eczema treatment plan provided to them by their healthcare provider.
  Family Dermatology Life Quality Index (FDLQI): Assess impact of the participant's eczema on the family's quality of life.
  Enrollment: Participants will complete FDLQI and PO-SCORAD.
  Week 1, 2, and 4: Participants will complete PO-SCORAD and AQ.
  Week 6: Participants will complete FDLQI, PO-SOCRAD, and AQ.
  Interventions: Behavioral: Patient reminders and accountability questionnaires
- No patient reminder/control (No Intervention): Participants in arm 2 are not sent text messages, and will not be asked to complete questionnaires 1, 2, and 4 weeks post enrollment. Participants will be asked to complete questionnaires during enrollment and 6 weeks post enrollment.
  Enrollment: Participants will complete FDLQI and PO-SCORAD.
  Week 6: Participants will complete FDLQI, PO-SOCRAD, and AQ.

INTERVENTIONS:
Behavioral: Patient reminders and accountability questionnaires — Participants who are assigned to the patient reminder arm will receive text messages 1, 2, and 4 weeks after enrollment. These text messages will encourage participants to adhere to the provided treatment plan, and ask participants to complete questionnaires to assess their adherence to treatment (in-house Adherence Questionnaire) and severity of eczema (PO-SCORAD) for that week.
  Arms: Patient reminder

SUMMARY:
Eczema is a chronic disease that requires long term and extensive treatment. However patient adherence to the treatment plans provided to them by their healthcare providers is poor. Frequent follow-up appointments have been demonstrated to improve treatment adherence, this may be due to patients feeling a sense of accountability which motivates them to adhere to their treatment. However, although frequent follow-up appointments are effective, they are not feasible. The goal of the Eczema Reminder and Accountability Program (ERAP) is to assess the effectiveness of a patient reminder system on patient adherence to treatment and the outcome of eczema. Participants will receive weekly/biweekly text messages that encourage them to adhere to their treatment plan, and asks them to assess the severity of their eczema and adherence to treatment for that week using questionnaires. Participants are then asked to send the completed questionnaires to Hamilton Allergy. Should the ERAP improve eczema outcome and treatment adherence, the goal is to use the ERAP as a virtual follow-up to reduce the need for frequent in-office follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Chronic atopic dermatitis.
* Age 0 to 16.

Exclusion Criteria:

-

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in severity of eczema | From date of randomization until 6 weeks post randomization. Time frame: 6 weeks.
  Participants will complete the Patient Oriented SCORAD (PO-SCORAD) to assess the severity of their eczema. Participants in arm 1 (reminders) will complete the PO-SCORAD on the date of randomization, and weeks 1, 2, 4, and 6 post randomization. Participants in arm 2 (no reminders) will complete the PO-SCORAD on the date of randomization and 6 weeks post randomization.
  To assess the impact of the ERAP on the outcome/severity of eczema, the change between the PO-SCORAD score from randomization and week 6 post randomization will be compared for arm 1 and arm 2.

SECONDARY OUTCOMES:
Treatment adherence | From 1 week post date of randomization until 6 weeks post date of randomization. Time frame: 5 weeks.
  Participants will complete the Adherence Questionnaire (AQ) to assess their adherence to the eczema treatment plan provided.
  Participants in arm 1 (reminders) will complete the AQ on weeks 1, 2, 4, and 6 post randomization.
  Participants in arm 2 (no reminders) will complete the AQ on week 6 post randomization.
  The AQ will be scored for week 6 post randomization and compared between arms 1 and 2 to determine the impact of the ERAP on treatment adherence.
Change in family quality of life | 6 weeks.
  To assess the impact of eczema on the family's quality of life, the participants' parents/guardians will be asked to complete the Family Dermatology Life Quality Index (FDLQI).
  Family members of participants in both arms 1 and 2 will be asked to complete the FDLQI on the date of randomization and 6 weeks post randomization.
  The change in FDLQI between the date of randomization and 6 weeks post randomization will be compared between arms 1 and 2 to assess the impact of the ERAP on the family's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Vince Wu, Principal Investigator — McMaster University
Locations (1):
- Hamilton Allergy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stalder JF, Barbarot S, Wollenberg A, Holm EA, De Raeve L, Seidenari S, Oranje A, Deleuran M, Cambazard F, Svensson A, Simon D, Benfeldt E, Reunala T, Mazereeuv J, Boralevi F, Kunz B, Misery L, Mortz CG, Darsow U, Gelmetti C, Diepgen T, Ring J, Moehrenschlager M, Gieler U, Taieb A; PO-SCORAD Investigators Group. Patient-Oriented SCORAD (PO-SCORAD): a new self-assessment scale in atopic dermatitis validated in Europe. Allergy. 2011 Aug;66(8):1114-21. doi: 10.1111/j.1398-9995.2011.02577.x. Epub 2011 Mar 18. PMID 21414011
- [Background] Basra MK, Sue-Ho R, Finlay AY. The Family Dermatology Life Quality Index: measuring the secondary impact of skin disease. Br J Dermatol. 2007 Mar;156(3):528-38. doi: 10.1111/j.1365-2133.2006.07617.x. PMID 17300244
- [Background] Bass AM, Anderson KL, Feldman SR. Interventions to Increase Treatment Adherence in Pediatric Atopic Dermatitis: A Systematic Review. J Clin Med. 2015 Jan 27;4(2):231-42. doi: 10.3390/jcm4020231. PMID 26239125